CLINICAL TRIAL: NCT05957601
Title: The Relationship Between the Parameters Affecting the Functionality of the Pelvic Floor and the Temporomandibular Joint
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Turkan Akbayrak, Prof. Dr., Hacettepe University
Other Study IDs: 14/07/2023
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Floor Disorders; Temporomandibular Joint Disorders
Keywords: pelvic floor; temporomandibular disorders
MeSH Terms: conditions — Pelvic Floor Disorders; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with pelvic floor dysfunction or healthy: All women who met the inclusion criteria, whether pelvic floor dysfunction or healthy, were included. If necessary, grouping can be done during statistics.
  Interventions: Other: No intervention was made as it was a descriptive epidemiological study.

INTERVENTIONS:
Other: No intervention was made as it was a descriptive epidemiological study. — No intervention was made as it was a descriptive epidemiological study.

SUMMARY:
The aim of our study is to examine the relationship between the parameters affecting the pelvic floor and temporomandibular joint (TMJ) functionality and to emphasize the necessity of investigating combined and coordinated exercise approaches in the treatment of dysfunctions that may occur in both specific regions. Our study, which is planned as an epidemiological research, will include 59 women between the ages of 20-50, who applied to the Istanbul Research and Training Hospital, Gynecology and Obstetrics Polyclinic, and volunteered to participate in the study. Assessments include pelvic floor dysfunction, pelvic floor muscle activation, sacroiliac joint mobility, pelvis position, and pain for pelvic floor functionality; temporomandibular joint dysfunction, masseter muscle activation, temporomandibular joint range of motion, position of the mandible and pain for temporomandibular joint funstionlaity; strength of the muscles located on the deep anterior line and thought to be related, flexibility, myofascial trigger points and depression level for mediating factors affecting functionality. After the data are completed, the Kolmogorov-Smirnov test will be applied to determine whether the data fit the normal distribution before starting the statistical analysis. Pearson Correlation test will be applied between dependent variables, independent variables and mediating factors in case the data show normal distribution, and Spearman Correlation test will be applied if it does not show normal distribution.

Significance value will be determined as p<0.05, correlation coefficient between variables r: 0-0.46 (weak); r: 0.5-0.74 (medium); r: will be interpreted as 0.75-1.0 (strong).

DETAILED DESCRIPTION:
It is known that there are postural changes in individuals with temporomandibular joint dysfunction (TMD). Although studies on this subject have focused mostly on the head, neck and shoulder regions, recent studies have shown that in addition to the opposite direction of head deviation and rectification in the thoracic region in individuals with TMD; It also indicates the presence of hyperlordosis in the lumbar region and posterior rotation of the pelvis. Similarly, Garstka et al. reported that unilateral sacroiliac joint locking was observed in individuals with clicking problems in temporomandibular joint (TMJ). Studies indicate that these effects of TMJ extending to the pelvic girdle occur through the facial pathways and that similar increases in symptoms in these regions are associated with emotional stress. A local change in a muscle segment first lengthens and shortens the muscles in close distance, and then acts on the other muscles on the fascial chain, thanks to the fascial pathways. The deep anterior fascial line starts from the sole of the foot and continues from the back of the leg bones to the inner side of the knee and thigh.While its main pathways pass in front of the hip joint, pelvis and lumbar spine, it proceeds with an alternate branch to the pelvic floor and the first lumbar spine. From the psoas-diaphragm space, it continues along several alternative pathways, covering the entire thorax and viscera, ending in both the neuro- and viscerocranium. Although the relationship of the TMJ with other structures on the connecting pathways has been the subject of many studies by looking at the fascial pathways of the deep anterior fascial line no study has been found that comprehensively examined the parameters of the TMJ and the pelvic floor. However, pelvic floor dysfunctions, urinary incontinence, faecal incontinence, pelvic organ prolapse, chronic pelvic pain, etc. It affects the psychology, physical condition, social life, family life, professional and sexual life of millions of women around the world. This study was planned because the etiology of dysfunctions of both regions is similar, they are located on the same fascial line, and although positive correlation results were obtained for other regions on the same fascial line, there was no previous study examining the relationship between TMJ and pelvic floor. In our study, we aim to emphasize the necessity of investigating combined and coordinated approaches in the prevention and treatment of dysfunctions that may occur in both specific regions by determining the relationship between the functionality of the pelvic floor and the TMJ and the factors affecting the relationship in women.

ELIGIBILITY:
Inclusion Criteria:

* having applied to the Istanbul Research and Training Hospital, Gynecology and Obstetrics Polyclinic,
* being literate
* being between 20-50 years old
* volunteering to participate in the study

Exclusion Criteria:

* pregnancy
* menopause
* having the cooperation problem
* history of active cancer
* urinary infection found during evaluation
* being in the period of menstruation at the time of assessment
* having a neurological, orthopedic or serious metabolic disease that may affect pelvic floor functions.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study was carried out only on women.
Study Population: All women with pelvic floor dysfunction or healthy who met the inclusion criteria were included in the study.
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pelvic floor dysfunction | Baseline
  Pelvic Floor Distress Inventory-20: There are 20 questions in total in the scale and these questions consist of 3 subfactors. According to whether they have the complaint or not, the participants say "no(0) or yes"; If the answers are yes, how much the complaint bothers the person will be graded as "insignificant (1), little (2), moderate (3), a lot (4)".
  The total score of the scale is between 0-300. The higher the score obtained as a result of this questionnaire, the higher the degree of complaint of pelvic floor dysfunction. Pelvic Organ Prolapse Quantification System: According to the hymen reference point, a total of 4 points will be measured: cervix, posterior fornix, anterior and posterior vaginal wall. According to the most distal point of the prolapse, Stage 0 (no prolapses); Stage I, Stage II, Stage III and Stage IV (complete eversion of the total length of the lower genital area).
Evaluation of temporomandibular joint dysfunction | Baseline
  Jaw Functional Limitation Scale - 20: Each item is scored between 0-10 on a scale consisting of 20 items. 0 = no restriction and 10 = severe restriction. The total score is between 0 and 200, and a high score indicates a high level of discomfort
Evaluation of pelvic floor muscle activation | Baseline
  Evaluation will be performed with the DuoBravo EMG device. The measurement is taken in the supine position, knees flexed 140 degrees, thighs and feet approximately 30 cm in order to completely relax the pelvic floor muscles, reduce the effect of gravity and eliminate auxiliary muscles such as hip adductors. open and the soles of the feet are in contact with the bed. The passive EMG electrode will be placed on the anterior surface of the thigh, and the active vaginal electrode will be placed intravaginally using a special probe for each patient. It will be clearly stated that when individuals are given the "relax" command, they should completely relax their pelvic floor muscles, and when the "muscle" command is given, they should only tighten the vaginal probe and pull it inward without contracting the hip, thigh and abdominal muscles and without holding their breath. The measurement will be repeated three times, the muscle activation response will be recorded in mV
Evaluation of masseter muscle activation | Baseline
  Evaluation will be performed with the DuoBravo EMG device. The active electrode will be placed on the most prominent point of the masseter muscle during isometric contraction, and the passive electrode will be placed on the nose. It will be clearly stated that when individuals are given the command "relax", they must completely relax their chewing muscles, and when the "muscle" command is given, they must perform a strong bite. The measurement will be repeated three times, the muscle activation response will be recorded in mV
Evaluation of sacroiliac joint mobility | Baseline
  Standing forward bending test: The physiotherapist will place both thumbs behind the participant, just below the Spina Iliaca Posterior Superior (SIPS). While the patient's knees are bent forward in extension, the physiotherapist will evaluate the asymmetry by following the movement with the thumbs. If one side is displaced more superiorly than the other, the test will be recorded as positive. For positive findings, Gillet's test will be done for confirmation.
Evaluation of temporomandibular range of motion | Baseline
  Evaluation will be carried out with a ruler. Painless mouth opening, maximum unaided mouth opening, maximum assisted mouth opening, right and left lateral movements will be measured with a ruler, values will be recorded in centimeters
Evaluation of pelvic pain | Baseline
  Pelvic Pain Impact Questionnaire: The questionnaire consists of 10 questions, but the first eight questions are scored.
  The range of points to be taken from the questionnaire varies between 1-32. The increase in the score value to be taken indicates that the effect of pelvic pain on the person also increases.
Evaluation of temporomandibular joint pain | Baseline
  Graded Chronic Pain Scale Version 2.0: The scoring of 6 items in the scale, which consists of 8 items in total, is made between 0 (no pain) and 10 (maximum pain), while the other 2 questions are evaluated by giving the number of days to the patient. A high score indicates a high level of discomfort.

SECONDARY OUTCOMES:
Evaluation of the strength of the muscles that are thought to be related and located on the Deep Anterior Facial Line | Baseline
  Evaluation will be performed with a LaFayette manual muscle strength measuring device for the tibialis posterior, adductors, iliopsoas, rectus abdominis, trapezius, and sternocleidomastoideus muscles. The measurement response will be recorded in pounds (Ibs)
Evaluation of flexibility | Baseline
  Sit-reach test: It will be used to evaluate the flexibility of hamstring muscles and trunk flexion. In the application of the test, the participant will be asked to sit on the test table with both knees extended, on a hard surface, and to reach for their hands and feet without bending their knees. The distance between the third finger of both hands and the tip of the test table will be measured with a ruler, and the value obtained will be recorded in centimeters.
  Trunk lateral flexion test: Participants will be asked to stand with their feet slightly open and parallel to each other, arms to the side of the trunk, and lateral flexion of the trunk. The distance in which the distal of the third finger of the patient was displaced was measured with the help of a tape measure and recorded in centimeters.
Evaluation of cervical range of motion | Baseline
  Evaluation will be performed with a goniometer as measurements of cervical flexion, extension, and right-left lateral flexion. The measurement response will be recorded in degrees
Evaluation of trigger points | Baseline
  Myofascial trigger points, which are frequently encountered in our body, will be evaluated by palpation (palpation will be done by pressing until the nail turns white, that is, with approximately 4 kilograms). Pain, twitching, and spread of pain over the palpable point are indicative of the presence of a trigger point, and if these symptoms are encountered, the presence of the trigger point will be recorded as "positive".
Evaluation of depression | Baseline
  Beck Depression Inventory: In the scale consisting of 21 questions, each question is scored between 0-3. The total score ranges from 0 to 63, and a high score indicates a high level of discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Akbayrak, Prof. Dr., Study Chair — Hacettepe University
Locations (1):
- Istanbul Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saito ET, Akashi PM, Sacco Ide C. Global body posture evaluation in patients with temporomandibular joint disorder. Clinics (Sao Paulo). 2009;64(1):35-9. doi: 10.1590/s1807-59322009000100007. PMID 19142549
- [Result] Garstka AA, Brzozka M, Bitenc-Jasiejko A, Ardan R, Gronwald H, Skomro P, Lietz-Kijak D. Cause-Effect Relationships between Painful TMD and Postural and Functional Changes in the Musculoskeletal System: A Preliminary Report. Pain Res Manag. 2022 Feb 28;2022:1429932. doi: 10.1155/2022/1429932. eCollection 2022. PMID 35265232
- [Result] Tim S, Mazur-Bialy AI. The Most Common Functional Disorders and Factors Affecting Female Pelvic Floor. Life (Basel). 2021 Dec 14;11(12):1397. doi: 10.3390/life11121397. PMID 34947928
- [Result] Toprak Celenay S, Akbayrak T, Kaya S, Ekici G, Beksac S. Validity and reliability of the Turkish version of the Pelvic Floor Distress Inventory-20. Int Urogynecol J. 2012 Aug;23(8):1123-7. doi: 10.1007/s00192-012-1729-8. Epub 2012 Mar 29. PMID 22456806
- [Result] Kaya S, Akbayrak T, Beksac S. Comparison of different treatment protocols in the treatment of idiopathic detrusor overactivity: a randomized controlled trial. Clin Rehabil. 2011 Apr;25(4):327-38. doi: 10.1177/0269215510385481. Epub 2010 Oct 13. PMID 20943711
- [Result] Ohrbach R, Larsson P, List T. The jaw functional limitation scale: development, reliability, and validity of 8-item and 20-item versions. J Orofac Pain. 2008 Summer;22(3):219-30. PMID 18780535
- [Result] Fridlund AJ, Cacioppo JT. Guidelines for human electromyographic research. Psychophysiology. 1986 Sep;23(5):567-89. doi: 10.1111/j.1469-8986.1986.tb00676.x. No abstract available. PMID 3809364
- [Result] Sahin D, Kaya Mutlu E, Sakar O, Ates G, Inan S, Taskiran H. The effect of the ischaemic compression technique on pain and functionality in temporomandibular disorders: A randomised clinical trial. J Oral Rehabil. 2021 May;48(5):531-541. doi: 10.1111/joor.13145. Epub 2021 Jan 21. PMID 33411952
- [Result] Alvarez DJ, Rockwell PG. Trigger points: diagnosis and management. Am Fam Physician. 2002 Feb 15;65(4):653-60. PMID 11871683